CLINICAL TRIAL: NCT06068400
Title: A Single-Arm, Single-Center Clinical Study to Evaluate the Safety and Efficacy of CAR-T in the Treatment of Multiple Myeloma
Brief Title: Clinical Study to Evaluate the Safety and Efficacy of CAR-T in the Treatment of Multiple Myeloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-CT-22-008
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma in Relapse
Keywords: Multiple Myeloma; BCMA; GPRC5D
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA/GPRC5D double CAR-T (Experimental): The study plans to enroll 40 subjects, with a sample size based on actual occurrence and a dosage of 3 × 106/kg ± 20%~1 × 107/kg ± 20% CAR positive T cells
  Interventions: Biological: BCMA/GPRC5D double CAR-T

INTERVENTIONS:
Biological: BCMA/GPRC5D double CAR-T — BCMA/GPRC5D double CAR-T is a new type CAR-T cells therapy for patients with Multiple Myeloma.

SUMMARY:
This is a single arm, single center clinical study evaluating the safety and efficacy of CAR-T treatment for multiple myeloma.

DETAILED DESCRIPTION:
This study is a single arm, single center study targeting patients with recurrent/refractory multiple myeloma (r/rMM). The study plans to enroll 40 subjects, with a sample size based on actual occurrence and a dosage of 3×106/kg±20%~1×107/kg ±20% CAR positive T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their guardians understand and voluntarily sign the informed consent form, and are expected to complete the follow-up examination and treatment of study procedures;
2. Aged 18-75 years, male or female;
3. According to IMWG diagnostic criteria, diagnosed with multiple myeloma;
4. Patients with documented multiple myeloma disease as relapsed refractory or primary refractory, defined as: a) relapsed refractory: no response to salvage therapy (no response defined as failure to achieve minimal response [MR] or disease progression on treatment), or disease progression within 60 days of the last treatment, or disease progression in patients who have achieved MR or above remission; b) primary refractory: never achieved MR or above response to any treatment, including never achieved MR or above remission, but M protein changes are not large, patients without evidence of clinical progression and patients who have primary refractory, progressed, and met the definition of progression.
5. the presence of measurable disease at screening as determined by any of the following criteria: serum monoclonal paraprotein (M-protein) level ≥ 1.0 g/dL or urine M-protein level ≥ 200 mg/24 hours; or diagnosis of light chain multiple myeloma without measurable disease in serum or urine: serum immunoglobulin free light chain ≥ 10 mg/dL and abnormal serum immunoglobulin κ/γ free light chain ratio; extramedullary measurable disease; the presence of tumor cells in the bone marrow as detected;
6. the patient has recovered from the toxicity of previous treatment, that is, CTCAE toxicity grade < 2 (unless the abnormality is tumor-related or judged by the investigator to be stable, it has little effect on safety or efficacy);
7. ECOG performance status score 0 to 2 and expected survival greater than 3 months;
8. Appropriate organ function:

alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal (ULN); aspartate aminotransferase (AST) ≤ 3 times the ULN; total bilirubin ≤ 1.5 times the ULN; Serum creatinine ≤ 1.5 times ULN, or creatinine clearance ≥ 30 mL/min (calculated by Cockcroft-Gault formula); Intraventricular oxygen saturation ≥ 92%; Left ventricular ejection fraction (LVEF) ≥ 45%, no pericardial effusion confirmed by echocardiography, no clinically significant electrocardiographic findings; no clinically significant pleural effusion; 9. venous access for collection can be established, no contraindications for leukocyte collection.

Exclusion Criteria:

1. Diagnosis or treatment of another invasive malignancy other than multiple myeloma within 3 years, with the following exceptions: malignancy treated with curative intent and no known active disease ≥ 3 years prior to enrollment; or adequately treated non-melanoma skin cancer with no evidence of disease;
2. previous anticancer therapy (prior to blood collection for CAR-T preparation) as follows: targeted therapy, epigenetic therapy, or investigational agent within 14 days or at least 5 half-lives (whichever is shorter), or invasive investigational medical devices; monoclonal antibody therapy within 21 days; proteasome inhibitor therapy within 14 days; immunomodulator therapy within 7 days; and radiotherapy within 14 days (except for bone marrow reserve with ≤ 5% field coverage);
3. Any hematopoietic stem cell transplantation within 2 months before screening;
4. History of central nervous system diseases;
5. known active central nervous system (CNS) involvement or clinical signs of meningeal involvement in multiple myeloma;
6. Waldenström macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal proteinopathy, and skin changes) or primary AL amyloidosis at screening;
7. Hepatitis B surface antigen (HBsAg) positive, or hepatitis B core antibody (HBcAb) positive and peripheral blood HBV DNA quantitative detection positive; hepatitis C virus (HCV) antibody positive; human immunodeficiency virus (HIV) antibody positive; cytomegalovirus (CMV) DNA detection positive; syphilis detection positive; Epstein-Barr virus DNA detection positive;
8. Patients with a history of severe allergy [a history of severe allergy is defined as a secondary or above allergic reaction, any of the following clinical manifestations occur when allergic reactions occur: airway obstruction (runny nose, cough, wheezing, dyspnea), tachycardia, hypotension, arrhythmia, gastrointestinal symptoms (nausea, vomiting), incontinence, laryngeal edema, bronchospasm, cyanosis, shock, respiratory, cardiac arrest] or known allergy to any of the active ingredients, excipients or murine products and xenogeneic proteins contained in this trial (including Qinglin regimen);
9. Patients with severe heart disease, including but not limited to severe arrhythmia, unstable angina pectoris, massive myocardial infarction, New York Heart Association class III or IV cardiac insufficiency, myocardial infarction ≤ 6 months before screening or coronary artery bypass grafting (CABG), a history of unexplained syncope and non-vasovagal or dehydration caused by, a history of severe non-ischemic cardiomyopathy, refractory hypertension (refractory hypertension is defined as: the use of reasonable tolerable adequate doses of ≥ 3 antihypertensive drugs (including diuretics) on the basis of lifestyle improvement for > 1 month of blood pressure is still not up to standard or taking ≥ 4 antihypertensive drugs blood pressure can be effectively controlled);
10. unstable systemic diseases judged by the investigator: including but not limited to severe liver, kidney or metabolic diseases requiring drug treatment;
11. Patients with acute/chronic graft-versus-host disease (GVHD) within 6 months before screening, or need to receive immunosuppressive agents for GVHD;
12. Patients with active autoimmune or inflammatory diseases of the nervous system (e.g., Guillain-Barre syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular disease (e.g., cerebral edema, posterior reversible encephalopathy syndrome (PRES));
13. Neoplastic emergencies (such as spinal cord compression, intestinal obstruction, leukostasis, tumor lysis syndrome, etc.) requiring emergency treatment before screening or reinfusion;
14. presence of uncontrollable bacterial, fungal, viral, or other infections requiring antibiotic therapy;
15. Hematopoietic cytokine drugs that have been transfused or have an effect on the hemogram of patients such as erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF), and granulocyte-macrophage colony-stimulating factor (GM-CSF) within 2 weeks of blood collection scheduled for CAR-T preparation at screening, and have an effect on cell preparation as judged by the investigator.
16. Receiving hormonal or immunosuppressive agents at screening within 2 weeks of blood collection scheduled for CAR-T preparation and having an effect on cell preparation as judged by the investigator.

1) Corticosteroids: subjects who are receiving systemic steroid therapy within 2 weeks of blood collection scheduled for CAR-T at screening and require chronic systemic steroid therapy during treatment as judged by the investigator (except for inhaled or topical use); and subjects who are receiving systemic steroid therapy within 72 hours before cell reinfusion (except for inhaled or topical use); 2) Immunosuppressants: subjects who are receiving immunosuppressive agents within 2 weeks of blood collection scheduled for CAR-T at screening; 17. Patients who have undergone major surgery (except diagnostic surgery and biopsy) within 4 weeks before Qinglin or plan to undergo major surgery during the study period, or whose surgical wounds have not completely healed before enrollment; 18. Patients who have received (attenuated) live viral vaccines within 4 weeks before screening; 19. patients with severe mental illness; 20. Alcoholics or those who have a history of drug abuse; 21. Pregnant or lactating women, and female subjects who plan to become pregnant within 2 years after cell reinfusion or male subjects whose partners plan to become pregnant within 2 years after cell reinfusion; 22. patients who have contraindications to any study procedure or have other medical conditions that may place them at unacceptable risk according to the investigator 's judgment and/or clinical criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Safety | Up to 2 years after BCMA/GPRC5D double CAR-T infusion
  Count the Incidence of adverse events
Changes in cytokine level | Up to 2 years after BCMA/GPRC5D double CAR-T infusion
  Calculate the change of cytokine level in peripheral blood by flow cytometry after CLL1 CAR-T infusion. Cytokines include IL-2、IL-6、IL-10、IFN-γ

SECONDARY OUTCOMES:
Complete response rate(CRR) | Up to 2 years after BCMA/GPRC5D double CAR-T infusion
  Proportion of subjects whose serum and urine immunofixation electrophoresis are negative, and there is no soft tissue plasma cell tumor, with bone marrow plasma cells<5%.
Strict complete response rate(SCRR) | Up to 2 years after BCMA/GPRC5D double CAR-T infusion
  Proportion of subjects who achieved complete response with normal FLC ratio and confirmed absence of clonal plasma cells in bone marrow by immunohistochemistry.
Very good partial response rate(VGPRR) | Up to 2 years after BCMA/GPRC5D double CAR-T infusion
  Proportion of subjects who detected serum and urine M protein in immunofixation, but did not detect it from electrophoresis; Or M protein decrease ≥ 90% and urine M protein<100 mg/24h.
Partial response rate(PRR) | Up to 2 years after BCMA/GPRC5D double CAR-T infusion
  Proportion of subjects who met the following requirements:
  1. A decrease of ≥ 50% in serum M protein and ≥ 90% or<200 mg/24h in urine M protein;
  2. If M protein in serum and urine cannot be detected, it is required to reduce the difference between affected and unaffected serum FLC by ≥ 50%;
  3. If M protein and serum FLC in serum and urine cannot be measured, and the baseline bone marrow plasma cell ratio is ≥ 30%, a reduction of ≥ 50% in the number of bone marrow plasma cells is required;
  4. In addition to the above criteria, if there is a baseline presence of soft tissue plasmocytoma, it is required that the sum of the maximum vertical diameter product (SPD) of the measurable lesion be reduced by ≥ 50%.
Minimal response rate(MRR) | Up to 2 years after BCMA/GPRC5D double CAR-T infusion
  Proportion of subjects whose serum M protein decreased by 25%~49% and 24-hour urine M protein decreased by 50%~89%; In addition to the above criteria, if there is a baseline presence of soft tissue plasmocytoma, a measurable reduction in lesion SPD of ≥ 50% is required.
Overall response rate(ORR) | Up to 2 years after BCMA/GPRC5D double CAR-T infusion
  Defined as the proportion of subjects who achieve sCR, CR, VGPR, and PR.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiao, MD, Principal Investigator — Shenzhen Qianhai Shekou Free Trade Zone Hospital
Locations (1):
- Shenzhen Qianhai Shekou Free Trade Zone Hospital, Shenzhen, Guangdong, China

REFERENCES:
- [Derived] Wei L, Xiao X, Jing X, Zheng Y, Sun X, Bai W, Li M, Luo M, Xiao Y. Case Report: Summary of multiple CAR-T expansions in anti-BCMA/GPRC5D bispecific CAR-T cell therapy for multiple myeloma. Front Immunol. 2025 Jun 6;16:1607778. doi: 10.3389/fimmu.2025.1607778. eCollection 2025. PMID 40547010